CLINICAL TRIAL: NCT02813239
Title: Dual Triggering With Gonadotropin-releasing Hormone Agonist and Standard Dose Human Chorionic Gonadotropin in Patients With a High Immature Oocyte Rate
Brief Title: Dual Triggering in Patients With a High Immature Oocyte Rate
Status: Completed | Type: Observational
Sponsor: IVI Madrid (Other)
Responsible Party: Principal Investigator, Juan A Garcia-Velasco, MD, IVI Madrid
Other Study IDs: 1408-MAD-058-JG
Record Dates: First submitted 2016-06-16; First posted 2016-06-24 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: INFERTILITY
Keywords: IVF; Dual trigger; GnRH agonist; hCG; mature oocytes
MeSH Terms: conditions — Infertility | interventions — Chorionic Gonadotropin; Gonadotropin-Releasing Hormone; Triptorelin Pamoate

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HCG triggering: Patients were scheduled by prescribing oral contraceptive (OC) for 12-16 days and recombinant FSH and/or highly purified u-hMG according to the patient's age, BMI, antral follicular count, AMH and previous responses to ovarian controlled stimulation. GnRH antagonist was added when at least one follicle reached 13 mm. Ovulation was induced by hCG when at least 2 follicles had a mean diameter of 17 mm.
  Interventions: Other: hCG
- HCG + GnRH agonist triggering: Patients were scheduled by prescribing oral contraceptive (OC) for 12-16 days and recombinant FSH and/or highly purified u-hMG according to the patient's age, BMI, antral follicular count, AMH and previous responses to ovarian controlled stimulation. GnRH antagonist was added when at least one follicle reached 13 mm. Ovulation was induced by hCG and GnRH agonist when at least 2 follicles had a mean diameter of 17 mm.
  Interventions: Other: hCG + GnRH agonist

INTERVENTIONS:
Other: hCG — Oocyte maturation with hCG
  Other Names: OVITRELLE (Merck Serono)
  Groups: HCG triggering
Other: hCG + GnRH agonist — Oocyte maturation with hCG + GnRH agonist
  Other Names: Ovitrelle (Merck Serono) + Decapeptyl (Ipsen Pharma)
  Groups: HCG + GnRH agonist triggering

SUMMARY:
In in vitro fertilization (IVF) cycles, even after adequate triggering, some patients present a high rate of immature oocytes retrieved after controlled ovarian stimulation. In vitro oocyte maturation is still an experimental technique, with poorer results than conventional IVF. For that reason improve in in vivo maturation could have a better impact on reproductive outcome.

DETAILED DESCRIPTION:
Investigators performed an observational study analyzing the difference in the percentage of mature oocytes retrieved in patients with more than 50% immature oocytes in a previous IVF cycle triggered with human chorionic gonadotropin (rhCG) compared to the rate of mature oocytes retrieved in subsequent cycles, triggered with both gonadotropin-releasing hormone agonist (GnRHa) and (hCG). The main outcome measure was the number and percentage of mature oocytes retrieved.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 18-30 kg/m2
* Male factor required for ICSI

Exclusion Criteria:

-

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women undergoing controlled ovarian stimulation with a high immature oocyte rate
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2014-11; Primary Completion 2014-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Metaphase II rate | 1 day
  Number of metaphase II among total of recovered oocytes

CONTACTS AND LOCATIONS:
Overall Officials: Juan Antonio Garcia Velasco, MD, Principal Investigator — IVI Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fatemi HM, Garcia-Velasco J. Avoiding ovarian hyperstimulation syndrome with the use of gonadotropin-releasing hormone agonist trigger. Fertil Steril. 2015 Apr;103(4):870-3. doi: 10.1016/j.fertnstert.2015.02.004. Epub 2015 Feb 24. PMID 25724740
- [Background] Kohls G, Ruiz F, Martinez M, Hauzman E, de la Fuente G, Pellicer A, Garcia-Velasco JA. Early progesterone cessation after in vitro fertilization/intracytoplasmic sperm injection: a randomized, controlled trial. Fertil Steril. 2012 Oct;98(4):858-62. doi: 10.1016/j.fertnstert.2012.05.046. Epub 2012 Jun 29. PMID 22749223